CLINICAL TRIAL: NCT07081750
Title: Development and Efficacy of a Dyadic Tailored Home-Based Activity Program for Mild-to-Moderate Dementia With Behavioral and Psychological Symptoms Post-Discharge: A Randomized Controlled Trial
Brief Title: Dyadic Tailored Home-Based Activity Program for Mild-to-Moderate Dementia Patients Post-Discharge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xiaozhen Fu, Graduate Researcher, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FY-EC-2025-304
Record Dates: First submitted 2025-07-06; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dementia
Keywords: dementia; behavioral and psychological symptoms; home-based; activity
MeSH Terms: conditions — Dementia; Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic tailored home-based activity program intervention (Experimental): （1） During hospitalization, caregivers receive health education on managing behavioral and psychological symptoms of dementia. Patient-caregiver dyads participate in structured ward activities to assess activity preferences and capabilities, forming the basis for co-developing individualized home activity plans with training for caregivers. （2） A customized home activity kit is provided at discharge. （3） Post-discharge, a 12-week tailored home intervention is implemented, using a patient-centered model with caregiver support. Caregivers record participation and behavioral responses, which inform dynamic adjustments to activity content, difficulty, and methods.
  Interventions: Behavioral: Dyadic tailored home-based activity program intervention
- Routine care (Active Comparator): Participants will receive routine care consisting of standard hospitalization treatment, basic caregiver education on behavioral and psychological symptoms of dementia (BPSD), routine discharge instructions (including general home activity recommendations without personalized intervention assessment, planning or implementation), and routine post-discharge follow-up for 12 weeks.
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: Dyadic tailored home-based activity program intervention — 1. During hospitalization, caregivers receive health education on managing behavioral and psychological symptoms of dementia. Patient-caregiver dyads participate in structured ward activities to assess activity preferences and capabilities, forming the basis for co-developing individualized home activity plans with training for caregivers.
  2. A customized home activity kit is provided at discharge.
  3. Post-discharge, a 12-week tailored home intervention is implemented, using a patient-centered model with caregiver support. Caregivers record participation and behavioral responses, which inform dynamic adjustments to activity content, difficulty, and methods.
  Arms: Dyadic tailored home-based activity program intervention
Other: Routine care — Participants will receive routine care consisting of standard hospitalization treatment, basic caregiver education on behavioral and psychological symptoms of dementia (BPSD), routine discharge instructions (including general home activity recommendations without personalized intervention assessment, planning or implementation), and routine post-discharge follow-up for 12 weeks.
  Arms: Routine care

SUMMARY:
This interventional study aims to evaluate the efficacy of a dyadic tailored home-based activity program in managing behavioral and psychological symptoms of dementia (BPSD) among home-dwelling people living with mild-to-moderate dementia post-discharge. The main question it aims to answer is:

Does the dyadic tailored home-based activity program significantly reduce BPSD in individuals with mild-to-moderate dementia after hospital discharge?

Researchers will compare people living with mild to moderate dementia who are receiving routine care to see if the dyadic tailored home-based activity program is effective for BPSD.

Participants will:

1. During hospitalization: People living with mild to moderate dementia and their caregivers receive health education on managing behavioral and psychological symptoms of dementia (BPSD); Participating activity sessions to assess individual preferences and functional activity capabilities, followed by co-designing a dyadic tailored home-based activity program.
2. After discharge: People living with mild to moderate dementia and their caregivers jointly receive a 12-week dyadic tailored home-based activity intervention at home.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Aged ≥60 years;
* ICD-10 diagnosed dementia with Clinician's Dementia Rating (CDR) scores of 1-2 (mild-to-moderate stage);
* Preserved basic verbal communication capacity;
* Exhibit at least one neuropsychiatric symptom (score ≥1 on any item) in the past month, as assessed by the Neuropsychiatric Inventory (NPI);
* Medically cleared for discharge with planned home-based care;
* Willing to provide written informed consent.

Caregivers:

* Aged ≥18 years;
* Designated primary caregiver (the individual spends the longest time caring for the patient each day);
* Committed to maintaining home caregiving responsibilities for at least 3 months post-discharge;
* Intact verbal communication skills;
* Possess basic operational proficiency with the WeChat application (capable of independently sending/receiving messages and conducting voice/video calls)
* Willing to provide written informed consent.

Exclusion Criteria:

Patients:

* Comorbid severe somatic diseases (e.g., malignant tumors, heart failure, physical disabilities) or psychiatric disorders;
* Severe visual or hearing impairment;
* Dementia caused by the following conditions: Central nervous system diseases (e.g., encephalitis, brain tumors, epilepsy, multiple sclerosis, Parkinson's disease); Nutritional/metabolic disorders (e.g., thyroid dysfunction, vitamin B12/folate deficiency); Substance or alcohol dependence; Other potential etiologies of secondary dementia;
* Severe physical or mental illness, extreme debilitation, long-term bedridden status, end-stage disease (with a life expectancy of less than six months), or an inability to cooperate with or tolerate the study;
* Currently participating in other medical research that may interfere with study outcomes.

Caregivers:

* Comorbid severe somatic diseases (e.g., malignant tumors, heart failure, physical disabilities) or psychiatric disorders;
* Severe visual or hearing impairment;
* Currently participating in other medical research that may interfere with study outcomes.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral and Psychological Symptoms of Dementia | Baseline and post-intervention (at the end of week 12)
  Assessment using the Neuropsychiatric Inventory (NPI) yields scores ranging from 0 to 144, with higher scores indicating more severe neuropsychiatric symptoms
Caregiver Distress of Behavioral and Psychological Symptoms of Dementia | Baseline and post-intervention (at the end of week 12)
  Assessment using the caregiver distress section of the Neuropsychiatric Inventory (NPI) yields scores ranging from 0 to 60, with higher scores indicating greater caregiver distress levels

SECONDARY OUTCOMES:
Cognitive Function of Dementia Patients | Baseline and post-intervention (at the end of week 12)
  Assessment using the cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-cog) yields scores ranging from 0 to 70, with higher scores indicating more severe cognitive impairment
Activities of Daily Living of Dementia Patients | Baseline and post-intervention (at the end of week 12)
  Assessment using the Activity of Daily Living (ADL) scale yields scores ranging from 20 to 80, with higher scores indicating more severe impairment in daily living activities.
Apathy of Dementia Patients | Baseline and post-intervention (at the end of week 12)
  Assessment using the Apathy Evaluation Scale-Informant version (AES-I) yields scores ranging from 18 to 72, with higher scores indicating more severe apathy symptoms
Agitation of Dementia Patients | Baseline and post-intervention (at the end of week 12)
  Assessment using the Cohen-Mansfield Agitation Inventory (CMAI) yields scores ranging from 29 to 203, with higher scores indicating more severe agitated behaviors
Quality of Life in Dementia | Baseline and post-intervention (at the end of week 12)
  Assessment using the Quality of Life-Alzheimer's Disease (QOL-AD) scale yields total scores ranging from 13 to 52, with higher scores indicating better quality of life
Caregiver Readiness for Hospital Discharge | Baseline
  Assessment using the Readiness for Hospital Discharge Scale-Caregivers (RHDS-C) yields total scores ranging from 0 to 220, with higher scores indicating better discharge readiness.
Caregiver Burden | Baseline and post-intervention (at the end of week 12)
  Assessment using the Caregiver Burden Inventory (CBI) yields scores ranging from 0 to 88, with a total score of <21 indicates no or mild burden, 21-39 suggests moderate burden, and ≥40 reflects severe burden.
Self Efficacy of Caregivers | Baseline and post-intervention (at the end of week 12)
  Assessment using the General Self-Efficacy Scale (GSES) yields scores ranging from 10 to 40, with higher scores indicating greater self-efficacy
Perceived Social Support of Caregivers | Baseline and post-intervention (at the end of week 12)
  Assessment using the Perceived Social Support Scale (PSSS) yields scores ranging from 12 to 84, with higher scores indicating greater perceived social support
Depression of Dementia Patients | Baseline and post-intervention (at the end of week 12)
  Assessment using the 24-item Hamilton Depression Scale (HAMD-24) yields total scores ranging from 0 to 78, with higher scores indicating more severe depressive symptoms. Specifically, scores <8 suggest no depression, 8-20 indicate possible depression, 21-35 confirm clinically significant depression, and >35 reflect severe depression
Depression of Caregivers | Baseline and post-intervention (at the end of week 12)
  Assessment using the 24-item Hamilton Depression Scale (HAMD-24) yields total scores ranging from 0 to 78, with higher scores indicating more severe depressive symptoms. Specifically, scores <8 suggest no depression, 8-20 indicate possible depression, 21-35 confirm clinically significant depression, and >35 reflect severe depression
Anxiety of Dementia Patients | Baseline and post-intervention (at the end of week 12)
  Assessment using the Hamilton Anxiety Scale (HAMA) yields total scores ranging from 0 to 56, with ≥29 indicating probable severe anxiety, ≥21 reflecting definite significant anxiety, ≥14 confirming anxiety presence, >7 suggesting possible anxiety, and <7 demonstrating no anxiety symptoms.
Anxiety of Caregivers | Baseline and post-intervention (at the end of week 12)
  Assessment using the Hamilton Anxiety Scale (HAMA) yields total scores ranging from 0 to 56, with ≥29 indicating probable severe anxiety, ≥21 reflecting definite significant anxiety, ≥14 confirming anxiety presence, >7 suggesting possible anxiety, and <7 demonstrating no anxiety symptoms.
Family Quality of Life in Dementia | Baseline and post-intervention (at the end of week 12)
  Assessment using the Family Quality of Life in Dementia Scale (FQOL-D) yields total scores ranging from 13 to 52, with higher scores indicating better family quality of life
Family Adaptability and Cohesion in Dementia | Baseline and post-intervention (at the end of week 12)
  Assessment was conducted using the Chinese Version of the Family Adaptability and Cohesion Scale, Second Edition (FACES II-CV), which comprises two subscales: Cohesion and Adaptability (15 items each, with subscale scores ranging from 15 to 75; higher scores indicate stronger family cohesion or adaptability
Number of Participants with Intervention-Related Adverse Events | Post-intervention (at the end of week 12)

OTHER OUTCOMES:
Number of caregivers with varying levels of satisfaction towards the intervention | Post-intervention (at the end of week 12)
Number of dementia patients with varying levels of satisfaction towards the intervention | Post-intervention (at the end of week 12)
Number of completed activity intervention sessions for dementia patients | Post-intervention (at the end of week 12)

IPD SHARING:
Plan to Share IPD: Yes